CLINICAL TRIAL: NCT00192166
Title: Trial to Assess Safety, Efficacy, Tolerability and Immunogenicity of Influenza Virus Vaccine, Administered Concomitantly With a Combination Live, Attenuated, Mumps, Measles, and Rubella Vaccine in Healthy Children Aged 11 - 24 Months
Brief Title: Trial to Assess Safety, Efficacy, Tolerability and Immunogenicity of Influenza Virus Vaccine, Liquid Formulation (CAIV-T), Administered Concomitantly With a Combination Live, Attenuated, Mumps, Measles, and Rubella Vaccine in Healthy Children Aged 11 - 24 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: D153-P522
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
- The primary objective of the study was to determine if intranasally administered influenza virus vaccine, CAIV-T), when administered concomitantly with a subcutaneously administered combination live, attenuated mumps, measles, and rubella (MMR) virus vaccine to children interferes with the immune responses.

DETAILED DESCRIPTION:
* The primary objective of the study was to determine if intranasally administered influenza virus vaccine, trivalent, types A and B, live, cold-adapted (CAIV-T), when administered concomitantly with a subcutaneously administered combination live, attenuated mumps, measles, and rubella (MMR) virus vaccine to children aged 11 to less than 24 months, interferes with the immune responses to the measles, mumps, and rubella components of the MMR vaccine.
* To compare the efficacy over one season against culture-confirmed influenza-illness caused by community-acquired subtypes antigenically similar to those contained in the vaccine, in children who are aged at least 11 months and less than 24 months at enrollment, between those who receive two doses of CAIV-T and those who receive placebo, each with concomitant administration of a combination live, attenuated MMR vaccine administered prior to the anticipated commencement of the influenza season.

ELIGIBILITY:
Inclusion Criteria:

* who were at least 11 months of age and less than 24 months of age at the time of first vaccination
* who were due to receive their first dose of combined measles, mumps, and rubella vaccine (MMR)
* who were in good health as determined by medical history, physical examination and clinical judgment
* whose parent(s)/legal guardian(s) provided written informed consent after the nature of the study was explained
* who, along with their parent(s)/legal guardian(s), were available for duration of the trial (approximately 8 months)
* whose parent(s)/legal guardian(s), could be reached by study staff for the post-vaccination contact (telephone, clinic or home visit)

Exclusion Criteria:

* whose parent(s)/legal guardian(s) were perceived to be unavailable or difficult to contact for evaluation or study visits during the study period
* who had any serious chronic disease (eg, with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease
* who had Down's syndrome or other known cytogenetic disorders who had a known or suspected disease of the immune system or those who received immunosuppressive therapy, including systemic corticosteroids. Subjects receiving high doses of systemic corticosteroids given daily or on alternate days, for 14 days or more, were excluded from vaccination until corticosteroid therapy was discontinued for at least one month. High doses were defined as 2 mg/kg/day or more of prednisolone or its equivalent, or 20 mg/day or more for children who weighed more than 10 kg.38
* who received, or were anticipated to receive, any blood products, including immunoglobulin, in the period from 6 months prior to vaccination through to the conclusion of the study
* for whom there was intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study had an immunosuppressed or an immunocompromised individual living in the same household
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational)
* who, at any time prior to entry into this study, received a dose of MMR vaccine or any of the individual components of the MMR vaccine (commercial or investigational)
* who were anticipated to receive a subsequent dose of MMR within 1 month after receipt of the second dose of CAIV-T or placebo
* with a documented history of hypersensitivity to egg or egg protein or any other components of CAIV-T or MMR
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the 2 weeks prior to vaccination or for which use is anticipated during the study
* with any medical conditions that in the opinion of the Investigator might have interfered with interpretation of the study results

Note: Pregnancy in any person who had regular contact with the subject was not a contraindication to the enrollment or ongoing participation of the subject in the study.

Ages: 11 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2002-10; Primary Completion 2003-03 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
All episodes of AOM, occurring during the influenza season, associated with a positive culture for influenza virus antigenically similar to those contained in the vaccine.

SECONDARY OUTCOMES:
The first episode during the influenza season of AOM associated with a positive culture for influenza virus; all episodes during the influenza season of AOM; all during the influenza season, of AOM associated with fever.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Chai-See Lum, Prof., Principal Investigator — University of Malaya Medical Centre
Locations (1):
- Respiratory Medicine Service, Singapore, Singapore